CLINICAL TRIAL: NCT02269111
Title: Quantitative High-Field Magnetic Resonance Imaging (MRI) for Assessing Brain Metastases
Brief Title: Quantitative MRI in Assessing Disease in Patients With Brain Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in PI and funding
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Albert Attia, Assistant Professor of Radiation Oncology; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC NEU1424; NCI-2014-01907 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC NEU1424 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Tumors Metastatic to Brain; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (hybrid MRI) (Experimental): Patients undergo hybrid 3 Tesla MRI examination that includes standard MRI sequences, DW-MRI, CEST, and combined DCE-MRI/DSC-MRI at baseline.
  Interventions: Procedure: diffusion-weighted magnetic resonance imaging; Procedure: chemical exchange saturation transfer magnetic resonance imaging; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Procedure: dynamic susceptibility contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Procedure: diffusion-weighted magnetic resonance imaging — Undergo DW-MRI
  Other Names: diffusion-weighted MRI
Procedure: chemical exchange saturation transfer magnetic resonance imaging — Undergo CEST-MRI
  Other Names: CEST MRI
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Undergo DCE-MRI
  Other Names: DCE-MRI
Procedure: dynamic susceptibility contrast-enhanced magnetic resonance imaging — Undergo DSC-MRI
  Other Names: DSC-MRI

SUMMARY:
This pilot clinical trial studies quantitative magnetic resonance imaging (MRI) at 3 Tesla in assessing disease in patients with tumors that have spread to the brain (brain metastases). In addition to routine care brain imaging of the brain, this study will include advanced multiparametric MRI sequences to measure vascular, cellular, and molecular properties of the tumor. Performing extra scans during MRI provides more information about the metastases and may better predict treatment response.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To correlate pre-treatment measures of biophysical parameters in metastases-obtained using advanced, quantitative MRI techniques in patients receiving standard-of-care (SOC) therapy for 1-4 brain metastases-with treatment-induced changes in lesion size, time-to-progression (TTP), and overall survival (OS).

OUTLINE:

Patients undergo hybrid 3 Tesla MRI examination that includes standard MRI sequences, diffusion-weighted (DW)-MRI, chemical exchange saturation transfer (CEST), and combined dynamic contrast enhanced (DCE)-MRI/dynamic susceptibility contrast (DSC)-MRI at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign an Institutional Review Board (IRB)-approved informed consent document
* Patients must have been diagnosed with one of the following:

  * Primary brain tumor (glioma, GBM etc); or
  * Up to 10 brain metastases
* Patients must have been diagnosed with 1-4 brain metastases
* At least one of the brain metastases must measure 5 mm (or more) in short axis diameter in the axial plane
* Patients must be scheduled to undergo standard brain cancer interventions:

  * Chemotherapy or targeted antiangiogenic therapy, in the case of primary brain tumor; or
  * Stereotaxic radiotherapy (SRS) or whole brain radiotherapy (WBRT), in the case of brain metastases.
* Patients must be scheduled to receive a 3-Tesla (3T) MRI exam as part of their standard of care (this exam will be modified to also include pulse sequences with are for research only)

Exclusion Criteria:

* Patients who have received previous treatment (chemotherapy or radiotherapy) for any brain tumor (primary or metastatic).
* Patients who are scheduled to receive a 1.5T MRI exam
* Patients incapable of giving informed written consent, due to mental disability, altered mental status, confusion, cognitive impairment, or psychiatric disorders.
* Patients scoring 14.5 or lower on the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) questionnaire will not be allowed on the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Volume transfer constant (Ktrans), as measured by DCE-MRI | Baseline
  The ability of pre-treatment estimates of Ktrans to predict objective tumor response by Response Evaluation Criteria in Solid Tumors or Macdonald criteria after therapy will be assessed using the proportional odds model.

SECONDARY OUTCOMES:
Amide proton transfer asymmetry (APTasym) as measured by CEST | Baseline
  Cox proportional hazards regression will be used to assess the association of APTasym with change in tumor size.
Apparent diffusion coefficient (ADC), as measured by DW-MRI | Baseline
  Cox proportional hazards regression will be used to assess the association of ADC with change in tumor size.
Extravascular extracellular volume fraction (Ve), as measured by DCE-MRI | Baseline
  Cox proportional hazards regression will be used to assess the association of Ve with change in tumor size.
Plasma volume fraction (Vp), as measured by DCE-MRI | Baseline
  Cox proportional hazards regression will be used to assess the association of Vp with change in tumor size.
Cerebral blood volume (CBV), as measured by DSC-MRI | Baseline
  Cox proportional hazards regression will be used to assess the association of CBV with change in tumor size.
Cerebral blood flow (CBF), as measured by DSC-MRI | Baseline
  Cox proportional hazards regression will be used to assess the association of CBF with change in tumor size.
Mean transit time (MTT), as measured by DSC-MRI | Baseline
  Cox proportional hazards regression will be used to assess the association of MTT with change in tumor size.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Attia, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/